CLINICAL TRIAL: NCT00656032
Title: Vitamin D, Insulin Resistance and Inflammation in ESRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080074
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: End Stage Renal Disease
Keywords: insulin resistance; end stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic; Insulin Resistance | interventions — paricalcitol; Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): SOC medication for treatment of renal osteodystrophy
  Interventions: Other: paricalcitol
- 2 (Active Comparator): alternate SOC medication for treatment of renal osteodystrophy
  Interventions: Other: cinacalcet

INTERVENTIONS:
Other: paricalcitol — 1 to 20 micrograms administered via IV; every other day, 3 days per week, for 8 weeks
  Other Names: zemplar
  Arms: 1
Other: cinacalcet — 0 to 180 mg administered orally every day for either 8 weeks or 16 weeks
  Other Names: sensipar
  Arms: 2

SUMMARY:
The broad goal of this study is to understand the mechanisms by which Vitamin D receptor activation leads to changes in insulin signaling in advanced uremia. We hypothesize that 1,25-Dihydroxyvitamin D3 deficiency due to advanced chronic kidney disease leads to insulin resistance and that administration of a vitamin D3 analog will restore insulin sensitivity in End Stage Renal Disease patients.

ELIGIBILITY:
Inclusion Criteria:

* CKD and receiving hemodialysis for ≥ 3months
* Kt/V ≥ 1.2
* ≥ 18 years of age
* Medically stable
* AVF or PTFE dialysis access
* No acute inflammatory disease within 4 weeks prior to the study
* On stable dose of Paricalcitol for 4 weeks prior to the study
* iPTH value between 150 - 1500 within the past 3 months
* Ca < 10.5
* PO4 < 10

Exclusion Criteria:

* Pregnancy
* Intolerance to the study medication
* Severe, unstable, active, or chronic inflammatory disease (active infection, active connective tissue disorder, active cancer, HIV, liver disease)
* Type 1 Diabetes mellitus
* Uncontrolled Type 2 Diabetes mellitus (HbA1c > 10)
* Hospitalization within 1 month prior to the study
* Malfunctioning arterial-venous vascular access (recirculation and/or blood flow < 250 ml/min)
* Presence of hemodialysis catheter
* Patients receiving steroids and/or other immunosuppressive agents (> 10 mg prednisone qd)
* BMI < 25 and > 45

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
An improvement in insulin sensitivity | 8 weeks

SECONDARY OUTCOMES:
A change in insulin signaling | 8 weeks
A decrease in concentration of plasma pro-inflammatory cytokines | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States